CLINICAL TRIAL: NCT03122184
Title: Positive Psychology for Acute Coronary Syndrome Patients: a Randomized, Controlled Pilot Trial
Brief Title: Positive Psychology for Acute Coronary Syndrome Patients
Acronym: PEACE-IV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jeff C. Huffman, MD, Associate Chief of Psychiatry for Clinical Services, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HL113272 (NIH)
Record Dates: First submitted 2017-04-06; First posted 2017-04-20 (Actual); Results first posted 2019-11-13 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: ACS - Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Psychology, Positive; Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Randomized, single-blinded, controlled trial
Who Masked: Outcomes Assessor
Masking Description: Participants and treating study staff will be aware of the patient's treatment condition. However, follow-up assessments will be performed by a study staff member that is masked to the participant's treatment condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Psychology + Motivational Interviewing (Experimental): Participants will complete weekly positive psychology exercises and will systematically set goals related to physical activity. Study trainers will review the positive psychology exercises on the phone each week and will use motivational interviewing techniques to facilitate goal setting.
  Interventions: Behavioral: Positive Psychology + Motivational Interviewing
- Motivational Interviewing Health Education (Active Comparator): Participants will speak on the telephone each week with a study trainer. During these calls, the trainer will provide education about a health behavior (physical activity, medication adherence, diet, stress reduction) and assign an activity related to one health behavior each week. Motivational interviewing techniques will be used throughout to facilitate health behavior changes.
  Interventions: Behavioral: Motivational Interviewing Health Education

INTERVENTIONS:
Behavioral: Positive Psychology + Motivational Interviewing — For the positive psychology portion of the intervention, the study trainer will (a) review the week's positive psychology exercise, (b) discuss the rationale of the next week's positive psychology exercise through a guided review of the positive psychology manual, and (c) assign the next week's positive psychology exercise. For the motivational interviewing portion, participants will (a) review their physical activity goal from the prior week, (b) discuss techniques for improving physical activity, and (c) set a physical activity goal for the next week. Study trainers will use motivational interviewing techniques to facilitate goal setting.
  Arms: Positive Psychology + Motivational Interviewing
Behavioral: Motivational Interviewing Health Education — Each week, participants will learn about a different health behavior topic related to cardiac health. They will also be introduced to motivational interviewing topics in concert with the health behavior education topics. The intervention is divided into five sections, focusing on five different important cardiac health-related topics (recovery from an acute cardiac illness, physical activity, a heart-healthy diet, medication adherence, and stress reduction).
  Arms: Motivational Interviewing Health Education

SUMMARY:
This is a randomized controlled pilot trial in approximately 50 acute coronary syndrome patients to determine if a 12 week, telephone-delivered, combined positive psychology-motivational interviewing intervention is feasible and more effective than a motivational interviewing health education program at improving health behaviors and other outcomes. The investigators hypothesize that the intervention will be associated with better mental and physical health outcomes and better health behavior adherence compared to the motivational interviewing health education program.

DETAILED DESCRIPTION:
The initial study visit will occur in-person two weeks after discharge from the hospital. Participants will meet with a member of the study staff (the study "trainer") and complete self-report questionnaires assessing health behavior adherence and mental and physical health. Then, participants will be randomized to receive the positive psychology + motivational interviewing or the motivational interviewing health education interventions. A study interventionist will provide a treatment manual specific to their condition, review the rationale for the initial exercise, and assign the first exercise. If the participant is in the positive psychology + motivational interviewing condition, the trainer will explain the rationale for both the positive psychology and goal-setting portions of the program, and will be assigned the first exercise. Similarly, if the participant is randomized into the motivational interviewing health education program, the interventionist will introduce them to the program and assign the first exercise. Participants in both groups will then be given an accelerometer, which they will be asked to wear for 7 days to ensure that they are comfortable with the device and that useable data can be obtained from the participant. Participants in both groups will then complete twelve 30-minute weekly phone sessions with a study trainer. The phone sessions primarily will include a review of the prior week's session content and a discussion of the rationale and assignment of the next week's exercise/assignment. Upon the completion of these calls, and again at a final follow-up timepoint at 24 weeks, a blinded member of the study staff will call participants to administer self-report outcome measures. Participants will also be asked to wear an accelerometer at each of these follow-up timepoints as an objective measure of physical activity, which they will return by mail to the study staff.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to Massachusetts General Hospital or Brigham and Women's Hospital inpatient units
* Diagnosis of acute coronary syndrome (using established criteria for myocardial infarction or unstable angina; confirmed via medical record and/or patient's treatment team)
* Age 18 or older
* Suboptimal adherence on MOS-SAS: Score < 15 OR Score = 15 with physical activity < 6

Exclusion Criteria:

* Cognitive deficits, assessed via a 6-item cognitive screen used to assess appropriate participation of medically ill patients in research studies.
* Medical conditions precluding interviews or likely to lead to death within 6 months, determined in consultation with the primary treatment team and cardiology co-investigator.
* Inability to perform moderate to vigorous physical activity, as defined by an inability to walk without aid of an assistive device such as a walker or cane, OR inability to walk at a steady pace for at least 5 minutes without stopping.
* Inability to communicate in English.
* Inability to participate in physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Huffman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 69 participants enrolled in the study but 22 either withdrew their consent or failed to attend their first in-person visit before randomization. Forty-seven individuals were randomized to a treatment condition.
Period: Overall Study
Arm/Group | Positive Psychology + Motivational Interviewing | Motivational Interviewing Health Education
Started | 24 | 23
Completed | 16 | 17
Not Completed | 8 | 6
Not completed — Lost to Follow-up | 4 | 6
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Terminated due to cognitive problem | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Positive Psychology + Motivational Interviewing | Motivational Interviewing Health Education | Total
Number analyzed (Participants) | 24 | 23 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 11 | 29
  >=65 years | 6 | 12 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 4 | 21
  Male | 7 | 19 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 23 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 24 | 19 | 43
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 23 | 47
Medication Adherence [Mean (Standard Deviation); unit: percentage of time] — Medication adherence was measured by the Self-Reported Medication Adherence (SRMA), a two-item self-report medication adherence scale measuring percentage of time (in 10% increments) patients report taking their heart medications in the past one and two weeks. Minimum: 0, Maximum:100. This measure was used at Baseline, Week 12, and Week 24.
  percentage of time | 95 (18) | 98 (4) | 97 (13)
Dietary Adherence [Mean (Standard Deviation); unit: score on a scale] — Measured by the MEDFICTS scale, a National Cholesterol Education Program-developed scale inquiring about saturated fat. Minimum= 0; Maximum= 216. Measure was used at Baseline, Week 12, and Week 24.
  score on a scale | 54.8 (27.4) | 55.4 (32.2) | 55.1 (29.5)
Positive Affect [Mean (Standard Deviation); unit: score on a scale] — The positive affect items on the Positive and Negative Affect Schedule (PANAS), a well-validated scale used in other intervention trials and in patients with medical illnesses, will be used to measure positive affect. (Range: 10-50). Higher scores indicate higher levels of positive affect. This measure was used at Baseline, Week 12, and Week 24.
  score on a scale | 28.5 (7.2) | 33.3 (6.3) | 30.9 (7.2)
Trait Optimism [Mean (Standard Deviation); unit: score on a scale] — Life Orientation Test-Revised is a well-validated 6-item instrument used to measure dispositional optimism. (Range: 0-24) Higher scores indicate higher levels of optimism. This measured was used at Baseline, Week 12, and Week 24.
  score on a scale | 16.1 (5.7) | 16.5 (4.6) | 16.3 (5.1)
State Optimisim [Mean (Standard Deviation); unit: score on a scale] — Measured by the State Optimism Scale developed by our team (SOM), which aims to capture the changeable nature of optimism based on time and situation. Minimum:7, Maximum:35. The higher number indicates a greater level of optimism. This measure was used at Baseline, Week 12, and Week 24.
  score on a scale | 25.8 (6.9) | 28.0 (5.4) | 26.9 (6.2)
HADS-A Score [Mean (Standard Deviation); unit: score on a scale] — The Hospital Anxiety and Depression Scale will be used to measure depression and anxiety. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients. (Range: 0-21) Higher scores indicate higher levels of anxiety. This measure was used at Baseline, Week 12, and Week 24.
  score on a scale | 5.5 (3.9) | 5.2 (4.0) | 5.3 (3.9)
HADS-D Score [Mean (Standard Deviation); unit: score on a scale] — The Hospital Anxiety and Depression Scale will be used to measure depression and anxiety. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients.(Range: 0-21). Higher scores indicate worse outcome (i.e. greater levels of depression). This measure was used at Baseline, Week 12, and Week 24.
  score on a scale | 4.0 (2.9) | 3.5 (2.4) | 3.7 (2.7)
Physical Function [Mean (Standard Deviation); unit: score on a scale] — Measured by the Duke Activity Status Index (DASI), a 12-item questionnaire that inquires about activities of daily living, basic physical activity, and more strenuous physical function to gauge overall functional capacity. Minimum: 0, Maximum: 58.2. Higher scores indicate greater levels of functional capacity. This measure was used at Baseline, Week 12, and Week 24.
  score on a scale | 37.3 (13.3) | 43.2 (13.9) | 40.2 (13.8)
SF-12 Scores (Physical) [Mean (Standard Deviation); unit: score on a scale] — The Medical Outcomes Study Short Form-12 (SF-12) will be used to measure quality of life. This is an instrument which has been used in multiple cardiac studies in the past. (SF-12 Mental Composite Score and Physical Composite Score Range: 0-100 each). Higher scores indicate higher level of health related QoL. This measure was used at Baseline, Week 12, and Week 24.
  score on a scale | 37.0 (7.0) | 40.0 (9.0) | 38.3 (8.0)
SF-12 Scores (Mental) [Mean (Standard Deviation); unit: score on a scale] — The Medical Outcomes Study Short Form-12 (SF-12) will be used to measure quality of life. This is an instrument which has been used in multiple cardiac studies in the past. (SF-12 Mental Composite Score and Physical Composite Score Range: 0-100 each). Higher scores indicate higher level of health related QoL. This measure was used at Baseline, Week 12, and Week 24.
  score on a scale | 46.9 (8.9) | 49.3 (8.0) | 48.1 (8.5)
Adherence to Health Behaviors [Mean (Standard Deviation); unit: score on a scale] — Three Medical Outcomes Study Specific Adherence Scale (MOS SAS) items assessing medication, diet, and exercise, will be measured individually and as a composite score. (Range: 3-18) Higher scores indicate better adherence to health behaviors. This measure was used at Baseline, Week 12, and Week 24.
  score on a scale | 9.9 (2.7) | 11.1 (2.6) | 10.5 (2.7)
Cardiac Symptoms [Mean (Standard Deviation); unit: score on a scale] — Measured by a checklist taken from the Women and Ischemia Syndrome Evaluation Study (WISE) to assess the presence and intensity of ten cardiac symptoms felt to best capture the range of symptoms experienced by ACS patients. Minimum: 0, Maximum: 30. Higher scores indicate greater levels of cardiac symptoms. This measure was used at Baseline, Week 12, and Week 24.
  score on a scale | 9.2 (5.2) | 8.5 (5.3) | 8.9 (5.2)
Physical Activity [Mean (Standard Deviation); unit: MET-minutes per week] — Measured by the self-report International Physical Activity Questionnaire (IPAQ). The measure assess the types of intensity of physical activity that people do as part of their daily lives. All activities are converted to multiples of resting energy expenditure (MET) minutes per week. This measure was used at Baseline, Week 12, and Week 24.
  MET-minutes per week | 2439.7 (5067.6) | 1809.8 (2266.8) | 2131.5 (3924.2)
Perceived Stress [Mean (Standard Deviation); unit: score on a scale] — Measured by the Perceived Stress Scale (PSS-4) measure. Minimum: 0, Maximum: 16. Higher scores indicate greater levels of stress. This measure was used at Baseline, Week 12, and Week 24.
  score on a scale | 5.7 (3.4) | 5.7 (2.7) | 5.7 (3.0)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of the PP-MI Based Health Behavior Intervention
Description: Feasibility will be measured by examining the number of completed exercises.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: exercises completed
Arm/Group | Positive Psychology + Motivational Interviewing
Number analyzed (Participants) | 24
exercises completed | 10.0 (3.9)

2. Primary Outcome: Acceptability of the PP-MI Exercises: Utility Score
Description: Participants will provide ratings of utility after each exercise, measured on a 10-point Likert scale (0=not at all helpful; 10=very helpful). Weekly utility ratings were averaged to provide an overall utility score of the exercises.
Time Frame: Weeks 1-12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Positive Psychology + Motivational Interviewing
Number analyzed (Participants) | 24
units on a scale
  Utility of the PP component | 8.0 (2.3)
  Utility of the MI component | 8.2 (2.2)

3. Primary Outcome: Acceptability of the PP-MI Exercises: Ease Score
Description: Participants will provide ratings of ease after each exercise, measured on a 10-point Likert scale (0=very difficult; 10=very easy). Weekly ratings were averaged to provide an overall ease of the exercises.
Time Frame: Weeks 1-12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Positive Psychology + Motivational Interviewing
Number analyzed (Participants) | 24
units on a scale
  Ease of the PP component | 8.3 (2.3)
  Ease of the MI component | 8.1 (2.4)

4. Secondary Outcome: Minutes of Moderate to Vigorous Physical Activity (Actigraph)
Description: ActiGraph GT3X+ step counters are validated as measures of physical activity and have been used in numerous studies of physical activity in patients with medical illness. In this trial, participants will wear the accelerometer for one week at 12 weeks, and another week at 24 weeks to assess the feasibility of doing so and to ensure adequate capture of physical activity. In our analysis, data on pre-ACS activity was collected using the International Physical Activity Questionnaire (IPAQ) to control for baseline activity.
Time Frame: MVPA at 12 weeks and 24 weeks
Population: Not everyone provided follow-up data at both time points.
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Positive Psychology + Motivational Interviewing | Motivational Interviewing Health Education
Number analyzed (Participants) | 18 | 16
minutes/day
  MVPA at 12-week: number analyzed (Participants) | 18 | 15
  MVPA at 12-week | 33.0 (19.0) | 23.2 (26.2)
  MVPA at 24-week: number analyzed (Participants) | 16 | 15
  MVPA at 24-week | 34.6 (22.9) | 18.1 (11.9)

5. Secondary Outcome: Change in Medication Adherence
Description: Measured by Self-Reported Medication Adherence (SRMA), a two-item self-report medication adherence scale measuring percentage of time (in 10% increments) patients report taking their heart medications in the past one and two weeks. Minimum: 0, Maximum:100. Change was calculated by subtracting the score at baseline from the score at 12 weeks and 24 weeks. Higher score indicates greater levels of medication adherence.
Time Frame: Change in score from Baseline to 12 weeks, 24 weeks
Population: Number of participants analyzed in Week 12 differs from that analyzed at Week 24 because not everyone provided data at both time points.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Positive Psychology + Motivational Interviewing | Motivational Interviewing Health Education
Number analyzed (Participants) | 20 | 21
percentage of time
  12 weeks: number analyzed (Participants) | 20 | 20
  12 weeks | 5 (2.2) | 5 (2.2)
  24 weeks: number analyzed (Participants) | 17 | 18
  24 weeks | 0 (0) | -6 (5.4)

6. Secondary Outcome: Change in Dietary Adherence
Description: Measured by the MEDFICTS scale, a National Cholesterol Education Program-developed scale inquiring about saturated fat. Minimum= 0; Maximum= 216. Change was calculated by subtracting the score at baseline from the score at 12 and 24 weeks. Higher scores indicate lower levels of dietary adherence.
Time Frame: Change in score from Baseline to 12 weeks, 24 weeks
Population: Number of participants analyzed in Week 12 differs from that analyzed at Week 24 because not everyone who provided data at both time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | Motivational Interviewing Health Education
Number analyzed (Participants) | 21 | 21
score on a scale
  12 weeks: number analyzed (Participants) | 20 | 20
  12 weeks | -2.8 (31.2) | -17.6 (21.5)
  24 weeks: number analyzed (Participants) | 18 | 17
  24 weeks | 2.1 (33.8) | -7.7 (25.6)

7. Secondary Outcome: Change in Positive Affect
Description: The positive affect items on the Positive and Negative Affect Schedule (PANAS), a well-validated scale used in other intervention trials and in patients with medical illnesses, will be used to measure positive affect. (Range: 10-50). Change was calculated by subtracting the score at baseline from the score at 12 and 24 weeks. Higher scores indicate higher levels of positive affect.
Time Frame: Change in score from Baseline to 12 weeks, 24 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | Motivational Interviewing Health Education
Number analyzed (Participants) | 20 | 20
score on a scale
  12 weeks | 8.8 (6.0) | 4.9 (6.5)
  24 weeks: number analyzed (Participants) | 17 | 17
  24 weeks | 9.5 (6.8) | 2.2 (6.6)

8. Secondary Outcome: Change in Trait Optimism
Description: Life Orientation Test-Revised is a well-validated 6-item instrument used to measure dispositional optimism. (Range: 0-24) Change was calculated by subtracting the score at baseline from the score at 12 and 24 weeks. Higher scores indicate higher levels of optimism.
Time Frame: Change in score from baseline to 12 week, 24 week
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | Motivational Interviewing Health Education
Number analyzed (Participants) | 20 | 20
score on a scale
  12 weeks | 2.2 (3.8) | 2.0 (5.3)
  24 weeks: number analyzed (Participants) | 17 | 17
  24 weeks | 1.7 (5.9) | 2.8 (3.8)

9. Secondary Outcome: Change in State Optimism
Description: Measured by the State Optimism Scale developed by our team (SOM), which aims to capture the changeable nature of optimism based on time and situation. Minimum:7, Maximum:35. The higher number indicates a greater level of optimism. Change was calculated by subtracting the score at baseline from the score at 12 and 24 weeks.
Time Frame: Change of score from Baseline to 12 weeks, 24 weeks
Population: Not all participants provided data at all follow-up points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | Motivational Interviewing Health Education
Number analyzed (Participants) | 20 | 19
score on a scale
  Change in SOM at 12 weeks | 5.3 (6.5) | -.1 (6.8)
  Change in SOM at 24 weeks: number analyzed (Participants) | 17 | 17
  Change in SOM at 24 weeks | 6.0 (7.1) | .6 (4.6)

10. Secondary Outcome: Changes in HADS-A Scores
Description: The Hospital Anxiety and Depression Scale will be used to measure depression and anxiety. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients. (Range: 0-21) Change was calculated by subtracting the score at baseline from the score at 12 and 24 weeks. Higher scores indicate higher levels of anxiety.
Time Frame: Change in score from Baseline to 12 week, 24 week
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | Motivational Interviewing Health Education
Number analyzed (Participants) | 20 | 19
score on a scale
  12 weeks | -2.8 (3.3) | -1.3 (2.8)
  24 weeks: number analyzed (Participants) | 17 | 17
  24 weeks | -2.3 (3.8) | -1.9 (2.0)

11. Secondary Outcome: Change in HADS-D Scores
Description: The Hospital Anxiety and Depression Scale will be used to measure depression and anxiety. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients.(Range: 0-21). Change was calculated by subtracting the score at baseline from the score at 12 and 24 weeks. Higher scores indicate worse outcome (i.e. greater levels of depression).
Time Frame: Change in score from Baseline to 12 week, 24 week
Population: We will use a random effects regression model with a random intercept for each participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | Motivational Interviewing Health Education
Number analyzed (Participants) | 20 | 19
score on a scale
  12 weeks | -1.8 (2.8) | .5 (2.5)
  24 weeks: number analyzed (Participants) | 17 | 17
  24 weeks | -1.5 (3.3) | -0.8 (2.2)

12. Secondary Outcome: Change in Physical Function
Description: Measured by the Duke Activity Status Index (DASI), a 12-item questionnaire that inquires about activities of daily living, basic physical activity, and more strenuous physical function to gauge overall functional capacity. Minimum: 0, Maximum: 58.2. Change was calculated by subtracting the score at baseline from the score at 12 and 24 weeks. Higher scores indicate greater levels of functional capacity.
Time Frame: Change of score from Baseline to 12 week, 24 week
Population: as for outcome 5
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | Motivational Interviewing Health Education
Number analyzed (Participants) | 20 | 20
score on a scale
  12 weeks: number analyzed (Participants) | 20 | 19
  12 weeks | 9.7 (11.7) | 4.4 (13.3)
  24 weeks: number analyzed (Participants) | 17 | 18
  24 weeks | 14.1 (13.0) | 4.9 (10.8)

13. Secondary Outcome: Change in SF-12 Scores (Physical)
Description: The Medical Outcomes Study Short Form-12 (SF-12) will be used to measure quality of life. This is an instrument which has been used in multiple cardiac studies in the past. (SF-12 Mental Composite Score and Physical Composite Score Range: 0-100 each). Change was calculated by subtracting the score at baseline from the score at 12 and 24 weeks. Higher scores indicate higher level of health related QoL.
Time Frame: Change of score from Baseline to 12 week, 24 week
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | Motivational Interviewing Health Education
Number analyzed (Participants) | 20 | 19
score on a scale
  12 weeks | 8.0 (8.0) | 7.2 (8.3)
  24 weeks: number analyzed (Participants) | 17 | 17
  24 weeks | 12.3 (7.4) | 6.8 (7.4)

14. Secondary Outcome: Change in SF-12 Scores (Mental)
Description: as for outcome 13
Time Frame: Change of score from baseline to 12 and 24 weeks.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | Motivational Interviewing Health Education
Number analyzed (Participants) | 20 | 19
score on a scale
  12 week | 8.8 (8.7) | 1.3 (5.8)
  24 week: number analyzed (Participants) | 17 | 17
  24 week | 6.3 (7.9) | 2.6 (4.8)

15. Secondary Outcome: Change in Adherence to Health Behaviors
Description: Three Medical Outcomes Study Specific Adherence Scale (MOS SAS) items assessing medication, diet, and exercise, will be measured individually and as a composite score. (Range: 3-18) Change was calculated by subtracting the score at baseline from the score at 12 and 24 weeks. Higher scores indicate better adherence to health behaviors.
Time Frame: Change of score from Baseline to 12 week, 24 week
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | Motivational Interviewing Health Education
Number analyzed (Participants) | 21 | 21
score on a scale
  12 weeks: number analyzed (Participants) | 20 | 20
  12 weeks | 4.9 (3.1) | 3.5 (2.7)
  24 weeks: number analyzed (Participants) | 18 | 18
  24 weeks | 4.4 (2.9) | 3.3 (3.4)

16. Secondary Outcome: Change in Cardiac Symptoms
Description: Measured by a checklist taken from the Women and Ischemia Syndrome Evaluation Study (WISE) to assess the presence and intensity of ten cardiac symptoms felt to best capture the range of symptoms experienced by ACS patients. Minimum: 0, Maximum: 30. Change was calculated by subtracting the score at baseline from the score at 12 and 24 weeks. Higher scores indicate greater levels of cardiac symptoms.
Time Frame: Change of score from Baseline to 12 week, 24 week
Population: Not all participants provided data at all follow-up points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | Motivational Interviewing Health Education
Number analyzed (Participants) | 20 | 19
score on a scale
  12 weeks | -6.6 (3.7) | -4.8 (4.4)
  24 weeks: number analyzed (Participants) | 17 | 17
  24 weeks | -6.6 (4.6) | -5.1 (4.3)

17. Secondary Outcome: Change in Physical Activity
Description: Measured by the self-report International Physical Activity Questionnaire (IPAQ). The measure asseses the types of intensity of physical activity that people do as part of their daily lives. All activities are converted to multiples of resting energy expenditure (MET) minutes per week. Change was calculated by subtracting the score at baseline from the score at 12 and 24 weeks.
Time Frame: Change of score from Baseline to 12 week, 24 week
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: MET-minutes per week
Arm/Group | Positive Psychology + Motivational Interviewing | Motivational Interviewing Health Education
Number analyzed (Participants) | 21 | 20
MET-minutes per week
  12 weeks: number analyzed (Participants) | 20 | 19
  12 weeks | 649.5 (1857.1) | 159.9 (4244.6)
  24 weeks: number analyzed (Participants) | 18 | 18
  24 weeks | -359.4 (1671.7) | -171.1 (2014.0)

18. Secondary Outcome: Change in Perceived Stress
Description: Measured by the Perceived Stress Scale (PSS-4) measure. Minimum: 0, Maximum: 16. Change was calculated by subtracting the score at baseline from the score at 12 and 24 weeks Higher scores indicate greater levels of stress.
Time Frame: Change of score from Baseline to 12 week, 24 week
Population: Not all participants provided data at all follow-up points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | Motivational Interviewing Health Education
Number analyzed (Participants) | 20 | 19
score on a scale
  12 weeks | -2.8 (3.0) | -1.4 (3.1)
  24 weeks: number analyzed (Participants) | 17 | 17
  24 weeks | -2.3 (3.0) | -2.5 (2.9)

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Adverse events are "any untoward or unfavorable medical occurrence in a human subject including any abnormal sign, symptom or disease...whether or not associated with the subject's participation in the research."
Arm/Group | Positive Psychology + Motivational Interviewing | Motivational Interviewing Health Education
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23
Serious Adverse Events (participants affected / at risk) | 11/24 | 11/23
Other Adverse Events (participants affected / at risk) | 7/24 | 6/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Positive Psychology + Motivational Interviewing (N=24) | Motivational Interviewing Health Education (N=23)
Unexpected chest and back pain (General disorders) | 1 (1) | 0 (0) — Patient admitted to hospital for chest and back pain.
Unexpected Coronary Artery Syndrome (Cardiac disorders) | 1 (1) | 2 (2) — Patient admitted to hospital for CAD.
Unexpected aneurysm (General disorders) | 0 (0) | 1 (1) — Patient admitted to hospital for nonruptured cerebral aneurysm.
Unexpected NSTEMI (Cardiac disorders) | 0 (0) | 1 (1) — Patient admitted to hospital for NSTEMI.
Unexpected hospital admission due to alt ms (General disorders) | 1 (1) | 0 (0) — Patient admitted to hospital for alt ms.
Unexpected fever (General disorders) | 1 (1) | 0 (0) — Patient admitted to hospital for fever.
Unexpected hypotension (Cardiac disorders) | 1 (1) | 0 (0) — Patient admitted to hospital for hypotension.
Unexpected sepsis (General disorders) | 1 (1) | 0 (0) — Patient admitted to hospital for sepsis.
Unexpected GI bleed (General disorders) | 1 (1) | 0 (0) — Patient admitted to hospital for GI bleed.
Unexpected calculus of gallbladder (General disorders) | 0 (0) | 1 (1) — Patient admitted to hospital for calculus of gallbladder without cholecystitis.
Unexpected melena (General disorders) | 0 (0) | 1 (1) — Patient admitted to hospital for melena.
Unexpected mass (General disorders) | 0 (0) | 1 (1) — Patient admitted to hospital for left renal mass.
Unexpected rectal bleeding (General disorders) | 1 (1) | 0 (0) — Patient admitted to hospital for Onc/Rectal bleeding.
Lymphoma (General disorders) | 1 (1) | 0 (0) — Patient admitted to hospital for lymphoma.
Unexpected A-FIB (General disorders) | 1 (1) | 1 (1) — Patient admitted to hospital for A-FIB
Unexpected Carpal Tunnel Syndrome (General disorders) | 0 (0) | 1 (2) — Patient admitted to FH for RIGHT CARPAL TUNNEL SYNDROME (SEVERE)
Unexpected eye damage (Eye disorders) | 1 (1) | 0 (0) — Patient admitted to hospital for Retinal detachment with single break, right eye.
Unexpected blood in stool (General disorders) | 0 (0) | 1 (1) — Patient admitted to hospital for blood in stool.
Unexpected malignant neoplasm of colon (General disorders) | 0 (0) | 1 (1) — Patient admitted to hospital for malignant neoplasm of descending colon.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Positive Psychology + Motivational Interviewing (N=24) | Motivational Interviewing Health Education (N=23)
Allergic reaction (General disorders) | 1 (1) | 0 (0) — Patient was admitted to the ED for an allergic reaction.
Stomach cramps and vomiting (General disorders) | 1 (1) | 0 (0) — Participant was admitted to ED for stomach cramps and vomiting.
Throat swelling (General disorders) | 1 (1) | 0 (0) — Participant was admitted to hospital for swelling in throat.
Abdominal pain (General disorders) | 1 (1) | 3 (5) — Participant was admitted to ED for abdominal pain.
Chest pain (Cardiac disorders) | 2 (2) | 1 (2) — Patient admitted to ED for chest pain
Chest discomfort (Cardiac disorders) | 1 (1) | 1 (2) — Patient admitted to ED for chest discomfort
Unexpected balance issues (General disorders) | 0 (0) | 1 (1) — Patient admitted to ED for unexpected balance issues

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT03122184/Prot_SAP_000.pdf